CLINICAL TRIAL: NCT04919447
Title: Study of the Efficacy and Safety of Cardiac Pacing of Different Sites
Brief Title: Clinical Study of LBBP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-675
Record Dates: First submitted 2021-06-07; First posted 2021-06-09 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Bradyarrhythmias; Heart Failure
MeSH Terms: conditions — Bradycardia; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: pacemaker implantation — cardiac pacing has been widely used in the treatment of bradyarrhythmias and heart failure, which can effectively improve the survival rate of patients.

SUMMARY:
At present, cardiac pacing has been widely used in the treatment of bradyarrhythmias and heart failure, which can effectively improve the survival rate of patients. With the rapid development of technology, you can choose to pace the heart in different parts. The atrium can choose the right atrial appendage, the atrial septum and the right ventricular side wall. The right ventricle can choose to be paced in the His bundle, right ventricular apex and ventricular septal outflow tract. The right ventricle can choose the pacing positions including left bundle branch pacing and left ventricular pacing via coronary vein. There are few studies comparing the long-term efficacy and safety of different pacing programs in daily practice. This study is to observe the short-term and long-term effects and safety of different parts of cardiac pacing, and compare the advantages and disadvantages of different parts of cardiac pacing.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received pacemaker implantation in the Second Hospital of Zhejiang Medical University by Pan Xiaohong and other surgeons.
* Patients who have the ability to understand the test and can cooperate with investigators.

Exclusion Criteria:

* Patients who unable to understand or unwilling to fill in informed consent forms or follow visitors

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: According to the current reports and the researcher's pacing implantation status, with an enrollment rate of 90% and a loss of follow-up rate of 10%, it is estimated that 600 cases were screened, 540 cases were selected, and about 500 cases were effective.
Sampling Method: Non-Probability Sample
Enrollment: 540 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Composite of Cardiovascular death, myocardial infarction, and stroke events | 60 months

CONTACTS AND LOCATIONS:
Locations (1):
- Xiaohong Pan, Hangzhou, Zhejiang, China